CLINICAL TRIAL: NCT00099814
Title: Clinical/Numerical Study of the Effects of Periodontal Ligament Stress Level on the Rate Bodily Tooth Movement
Brief Title: Periodontal Ligament Stress Level and Tooth Movement
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Joanne Lafrance, research assistant, University of Alberta, Graduate Orthodontic Program
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: GOP-UA-CT-01
Record Dates: First submitted 2004-12-21; First posted 2004-12-21 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Malocclusion, Angle Class III
Keywords: tooth movement; orthodontics; force; humans; clinical trial
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Two different loop designs which deliver distinctive forces

SUMMARY:
Orthodontic treatment requires application of force systems to individual teeth or groups of teeth, which results in a cellular response with periodontal ligament (PDL) and alveolar bone remodeling. The forces applied must be of sufficient magnitude and duration to exceed the normal physiologic threshold associated with daily oral function. Excessive force levels will result in areas of tissue necrosis with delayed tooth movement and increased risk of root resorption. Although orthodontic tooth movement is achieved in a large segment of the population, the optimum force level has not been defined. The optimum force for tooth movement depends on individual root geometry as well as biologic characteristics of surrounding tissue including bone density, periodontal thickness, and fluid dynamics.

Because experimental and clinical techniques are generally limited to known complex force systems, biomechanical modeling has become a necessity. Such models must be validated with well-controlled clinical studies that evaluate orthodontic tooth movement over an extended distance. The ultimate goal would be development of a computer simulation model to predict tooth movement in the clinical setting.

The primary objective of this study is to test controlled clinical data with a biomechanical model of the tooth and supporting tissues for distal movement of the human maxillary canine tooth (of known root geometry) in response to various 3D force systems that produce different levels of stress in the supporting tissues. Secondary objectives include evaluation of rate of bodily tooth canine movement with two known compressive stress levels (13 and 22 kPa), evaluation of three different reference systems to measure rate of tooth movement, and evaluation of an implant placed in the roof of the mouth (palatal implant) for orthodontic anchorage in adolescent patients.

The rate of translation (bodily) tooth movement of the maxillary canine tooth will be significantly greater with 22kPa compared to 13kPa compressive stress applied to the periodontal ligament, and this difference can be predicted by appropriate mathematical/numerical models of the tooth and supporting tissues.

DETAILED DESCRIPTION:
The patients will be drawn from those recruited for the Graduate Orthodontic Graduate Program. Clinical academic staff will examine approximately 500 patients seeking orthodontic care. Patients are categorized by malocclusion type and placed into a patient pool from which some cases are selected for treatment based on the program teaching and research needs. Each year approximately 50% of patients seeking care are ultimately accepted. Treatment is provided at fees that are approximately 60% of those charged in private practice.

Patients who meet the selection criteria for this study will be randomly selected from the University of Alberta Graduate Orthodontic Graduate Clinic patient pool. Upper 1st premolar teeth will be extracted and full fixed orthodontic appliances (Ormco Orthos prescription) will be placed. After the initial alignment and leveling phase is completed the retraction phase will begin. Non-steroidal anti-inflammatory agents will be avoided; only extra strength Tylenol will be prescribed as necessary for any momentary pain or discomfort. Maximum posterior anchorage will be attained through a palatal implant (Straumann) according to the protocol described by Papadakis. The implants will be also used as three-dimensional movement reference points. Other reference systems to be used include the palatal ruggae and occlusal templates. The cuspid retraction force delivery mechanisms will consist of customized activated stainless steel T-loops designed to generate the required forces on the bracket. Approximate compressive stress (based on approximate root surface area) of 13 kPa and 22 kPa will be applied on the distal aspect of the cuspids. The design will be a split-mouth study in which both levels of stress will be applied in each patient. The side to which the higher and lower stress levels are applied will be randomized. This design will allow for inter and intra-patient comparisons since each patient will see both stress levels. After the initial activation the subjects will be seen at day 1, 3, 17 and thereafter at 4-week intervals until the space between the cuspid and second bicuspid is completely closed. In the initial activation session and each of the follow-up sessions, maxillary impressions and appliance adjustments to apply the desired force will be made. At each clinical visit impressions will be made of the activated T-loop and the teeth. The geometry of the T-loop will be measured from the impressions which will allow for the applied force to be calculated using a numerical method developed by Raboud. The impression of the teeth will be used to construct the occlusal templates required to measure tooth movement.

Tooth mobility change during the orthodontic tooth movement will be monitored by means of the Periotest measuring device. CT volumetric scans with the NewTom machine will be made just before placement of the implant to ensure adequate palatal bone volume. Extra CT volumetric scans will be repeated in the middle of the retraction period (based on the space to be closed) and at the end of the space closure. The CT volumetric scan images will also be used to determine alveolar bone density, changes in root geometry for calculation of root surface area and center of resistance. The CT volumetric scans will also be used to determine alveolar bone density, change in root geometry (root resorption) and to assess movement of the cuspid in relation to other maxillary structures. The series of models from each subject and a 3-axis measuring system (MicroVal) will be used to measure tooth position changes relative to the 3 reference systems.

At the completion of cuspid retraction, the balance of the required orthodontic treatment will continue. The palatal implant will be retrieved and orthodontic retention delivered. Data gathered in the patient study will be utilized to validate the biomechanical model.

Biomechanical Modeling:

There will be two separate biomechanical tooth models developed. The first will be a parametric three dimensional model of the tooth and supporting tissues which will allow for variable biological properties of the tooth, PDL and alveolar bone. This model allows the inputs to be patient specific for both the force systems applied and the individual biological parameters. The three dimensional force systems that are applied to the tooth will be calculated using the numerical method described by Raboud and the measured geometry of the T-loop. The Finite Element Model (FEM) of the tooth and supporting tissue and the applied force system will allow for an improved description of the stress fields in the tissues, in particular the PDL. This improved stress field will be compared to the resulting bodily tooth movement. In order to compare the results from the biomechanical model and the clinical study it is important that the posterior segment does not move. The palatal implant is to ensure the absolute anchorage required.

As previously mentioned, the accuracy of the FEM model is dependant upon the input parameters. Consequently, there will be a two dimensional dynamic model of the tooth response to a mechanical impact. This will model instruments such as the Periotest® which is designed to measure impact response. Since the tooth response is governed by the characteristics of the periodontal ligament, analysis of the raw signal obtained from the Periotest® will allow for the mechanical properties of the PDL to be evaluated during the retraction.

Statistical Analysis:

The final mean rate of tooth movement between the two force levels will be compared through the Independent Samples T Test. To evaluate significant changes of the tooth movement in the distinctive time intervals, a repeated measure ANOVA will be used. If the underlying assumptions for both methods are not satisfied, then the non-parametric alternative will be considered (U Mann-Whitney Test).

ELIGIBILITY:
Inclusion Criteria:

* Female adolescent (12-16 years old) orthodontic patients requiring upper first premolars extractions for overjet reduction.
* Participants will be healthy and not taking any medications.
* All participants will have healthy periodontal tissues and good oral hygiene.

Exclusion Criteria:

* Patients with medical contraindication for placement of a palatal implant.
* All candidates who admit to tobacco utilization will be excluded.
* Patients requiring lower dental extractions will also be excluded.
* Pregnant patients or patients planning pregnancy will be excluded.

Ages: 12 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20
Dates: Start 2004-03; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Rate of space closure

CONTACTS AND LOCATIONS:
Locations (1):
- Orthodontic Clinic - Department of Dentistry - University of Alberta, Edmonton, Alberta, Canada